CLINICAL TRIAL: NCT04773184
Title: Improving Clinical and Instrumental Diagnostic Standards in Dysphagia.
Brief Title: Improving Diagnostic Standards in Dysphagia
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202003199; OCR40105 (Other: UF OnCore)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Dysphagia
Keywords: Dysphagia; Peak Cough Flow (PCF); Swallowing; Respiration
MeSH Terms: conditions — Deglutition Disorders; Respiratory Aspiration | interventions — Fees and Charges; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy adults: 132 individuals with no history of swallowing impairment or any health conditions known to impact swallowing function will be included in this study to serve as a comparative control group or reference standard group here and in future studies.
  Interventions: Procedure: Fiberoptic Endoscopic Evaluation of Swallowing; Procedure: Videofluoroscopic Swallowing Study; Procedure: Voluntary Peak Cough Flow Testing; Procedure: Iowa Oral Performance Instrument; Procedure: Capsaicin Challenge; Procedure: Pulmonary Function Testing; Other: Voicing Tasks
- Adults at risk for swallowing impairment.: 132 individuals with an underlying condition documented to lead to dysphagia will be enrolled in this study. 2) Confirmed medical diagnosis associated with an increased risk of dysphagia including but are not limited to: head and neck cancer, neurologic (e.g., stroke, traumatic brain impairment), neurodegenerative (e.g., Parkinson's disease, amyotrophic lateral sclerosis), neuromuscular disorders (e.g., myotonic dystrophy, Pompe disease, inclusion body myositis) rheumatologic diseases (e.g., dermatomyositis, inclusion body myositis, scleroderma), chronic respiratory illnesses (e.g., chronic obstructive pulmonary disease), structural (e.g., mass or trauma to the upper aerodigestive tract) and iatrogenic conditions (e.g., post-surgical such as anterior cervical discectomy/fusion or cardiac, post-radiation treatment to the upper aerodigestive tract).
  Interventions: Procedure: Fiberoptic Endoscopic Evaluation of Swallowing; Procedure: Videofluoroscopic Swallowing Study; Procedure: Voluntary Peak Cough Flow Testing; Procedure: Iowa Oral Performance Instrument; Procedure: Capsaicin Challenge; Procedure: Pulmonary Function Testing; Other: Voicing Tasks

INTERVENTIONS:
Procedure: Fiberoptic Endoscopic Evaluation of Swallowing — This procedure involves inserting a flexible laryngoscope that contains a light source and video camera on the end through the open passage of the nose towards the back of the throat in order to visualize the swallowing mechanism.
  Other Names: (FEES)
Procedure: Videofluoroscopic Swallowing Study — Videofluoroscopic swallowing study will be performed to measure oropharyngeal swallowing. This is like a moving x-ray of the swallow.
Procedure: Voluntary Peak Cough Flow Testing — Voluntary peak cough flow testing will be performed to determine the peak expiratory flow (PEF) and volume of air expelled (FEV1) during voluntary coughing.
Procedure: Iowa Oral Performance Instrument — The Iowa Oral Performance Instrument (IOPI) is a device that measures the peak pressure performance of lingual strength and endurance via the action of a bulb placed on the hard palate.
Procedure: Capsaicin Challenge — A capsaicin challenge with three randomized blocks of 0, 50, 100, 200, and 500 μM capsaicin. The capsaicin will be dissolved in a vehicle solution consisting of 80% physiological saline, and 20% ethanol. Participants will be given the instruction "cough if you need to" prior to capsaicin delivery.The solution will be administered automatically upon detection of an inspired breath and there will be a minimum of one minute between each trial. This is to test the reflexive cough testing for upper airway sensitivity and motor thresholds.
  Other Names: Reflexive Cough Testing
Procedure: Pulmonary Function Testing — Pulmonary Function testing will be performed using conventional methods and will include the following outcomes: forced vital capacity (FVC), maximum inspiratory pressure (MIP), and maximum expiratory pressure (MEP) expressed as a percentage of predicted values.
Other: Voicing Tasks — Voicing tasks will be completed to assess vocal ability.

SUMMARY:
The purpose of this research is to understand the normal function of swallowing and respiratory muscles in order to establish normal parameters. This will allow us to compare normal physiology and function of swallowing and breathing muscles to people with a medical history that would put them at risk for a swallowing problem. Our goal is to identify the best tests that can be quickly and easily administered to accurately detect swallowing impairment in adults. Involvement is limited to a single 2-hour evaluation.

DETAILED DESCRIPTION:
The purpose of this research is to understand the normal function of swallowing and respiratory muscles in order to establish normal parameters. It will take approximately 90-120 minutes to complete. During this examination, you will have respiratory testing, cough testing, lingual testing, voice testing, and will be asked to fill out some surveys. We will then complete the swallowing test that uses both a moving x-ray and a small camera will be inserted into the open passage of your nose to the back of your throat to watch your swallow and look at your vocal folds (voice box). This will allow us to compare normal physiology and function of swallowing and breathing muscles to people with a medical history that would put them at risk for a swallowing problem. Our goal is to identify the best tests that can be quickly and easily administered to accurately detect swallowing impairment in adults. Your involvement is limited to a single 2-hour evaluation.

ELIGIBILITY:
Healthy Cohort:

132 individuals with no history of swallowing impairment or any health conditions known to impact swallowing function will be included in this study to serve as a comparative control group or reference standard group here and in future studies.

Inclusion criteria:

1. Adults aged 18-90.
2. No history of stroke, head and neck cancer or other disorder that might contribute to a swallowing impairment.
3. No COVID-19 symptoms within the past 14 days, nor has been around someone testing positive for COVID-19 in the past 14 days.
4. Not pregnant.
5. No allergies to barium.

Exclusion criteria:

1. Individuals under the age of 18 or over the age of 90.
2. History of stroke, head and neck cancer or other disorder that might contribute to a swallowing impairment.
3. Within the past 14 days, individuals with COVID-19 symptoms or a positive COVID-19 test, or who have been exposed to someone with confirmed COVID-19.
4. Pregnant women.
5. Individuals with allergies to barium.

Disordered Cohort:

132 individuals with an underlying condition documented to lead to dysphagia will be enrolled in this study.

Inclusion criteria:

1. Adult participants aged between 18 and 90 years.
2. Confirmed medical diagnosis associated with an increased risk of dysphagia including but are not limited to: head and neck cancer, neurologic (e.g., stroke, traumatic brain impairment), neurodegenerative (e.g., Parkinson's disease, amyotrophic lateral sclerosis), neuromuscular disorders (e.g., myotonic dystrophy, Pompe disease, inclusion body myositis) rheumatologic diseases (e.g., dermatomyositis, inclusion body myositis, scleroderma), chronic respiratory illnesses (e.g., chronic obstructive pulmonary disease), structural (e.g., mass or trauma to the upper aerodigestive tract) and iatrogenic conditions (e.g., post-surgical such as anterior cervical discectomy/fusion or cardiac, post-radiation treatment to the upper aerodigestive tract).
3. No COVID-19 symptoms within the past 14 days, nor has been around someone testing positive for COVID-19 in the past 14 days.
4. Not Pregnant.
5. No allergies to barium.

Exclusion criteria:

1. Individuals under the age of 18 or over the age of 90
2. Within the past 14 days, individuals with COVID-19 symptoms or a positive COVID-19 test, or who have been exposed to someone with confirmed COVID-19.
3. Pregnant women.
4. Individuals with allergies to barium.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Cohort:
  132 individuals with no history of swallowing impairment or any health conditions known to impact swallowing function will be included in this study to serve as a comparative control group or reference standard group here and in future studies.
  Disordered Cohort:
  132 individuals with an underlying condition documented to lead to dysphagia will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale | Baseline
  Validated swallowing safety measurement that is an eight-point ordinal scale to indicate the depth of airway invasion during swallowing and the associated response. A minimum score of 1 would be no airway invasion, to a maximum score of 8 being airway invasion with no effort to expel the tracheal matter. Therefore, the lower the score, the better the outcome.
Yale Residue Severity Rating Scale | Baseline
  Validated measure of swallowing efficiency using a validated anatomically defined and image-based assessment of post-swallow pharyngeal residue severity. Clinical uses include accurate classification of vallecula and pyriform sinus residue severity patterns as none, trace, mild, moderate, or severe for diagnostic purposes, determination of functional therapeutic change, and precise dissemination of shared information.
Vocal Fold Mobility Impairment | Baseline
  During a Fiberoptic Endoscopic Evaluation of Swallowing (FEES), the vocal folds will be visualized using a small camera passed through the open nasal passage. The patient will be asked to make a series of vocal tasks so that we can visualize their movement, any immobility will be notated.
Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) | Baseline
  5-point ordinal scale used to rate both the safety and efficiency of swallowing trials. For efficiency, the minimal score of 0 means residue is less than 10%, the maximal score of 4 means there is more than 90% of residue across trials. For safety a minimal score of 0 means no airway invasion, and a maximal score of 4 means there was chronic and gross amounts of food or liquids that were aspirated. Therefore, the lower the scores, the better the outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Plowman, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
None at this time